CLINICAL TRIAL: NCT03615482
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 When Administered Concomitantly With Influenza Vaccine in Healthy Adults 50 Years of Age or Older (PNEU-FLU)
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 When Administered Concomitantly With Influenza Vaccine in Healthy Adults 50 Years of Age or Older (V114-021/PNEU-FLU)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V114-021; V114-021 (Other: Merck Protocol Number)
Record Dates: First submitted 2018-07-31; First posted 2018-08-03 (Actual); Results first posted 2020-06-29 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Concomitant Vaccination (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V114 and a single 0.5 mL IM injection of QIV on Day 1 and a single 0.5 mL injection of placebo on Day 30
  Interventions: Biological: V114; Biological: QIV; Biological: Matching Placebo for V114
- Non-concomitant Vaccination (Experimental): Participants will receive a single 0.5 mL IM injection of QIV and a single 0.5 mL IM injection of placebo on Day 1 and a single 0.5 mL injection of V114 on Day 30
  Interventions: Biological: V114; Biological: QIV; Biological: Matching Placebo for V114

INTERVENTIONS:
Biological: V114 — Single 0.5 mL injection
Biological: QIV — Single 0.5 mL injection
  Other Names: Quadrivalent influenza vaccine (seasonal inactivated); Fluarix Quadrivalent (Influenza Vaccine)
Biological: Matching Placebo for V114 — Single 0.5 mL injection

SUMMARY:
This study was designed to evaluate the safety and tolerability of a single dose of V114 when administered concomitantly and non-concomitantly (i.e., 30 days after) with influenza vaccine. It also evaluated whether V114 can be administered concomitantly with influenza vaccine without impairing the antibody response to the 15 serotypes contained in V114 and to the 4 influenza viruses contained in the seasonal inactivated quadrivalent influenza vaccine (QIV). The primary hypotheses state that immune responses to V114 and to QIV are non-inferior when administered concomitantly as compared with non-concomitant administration as measured by serotype-specific opsonophagocytic activity (OPA) and hemagglutination inhibition (HAI) geometric mean titers (GMTs) at 30 days postvaccination. This study will also contribute to the overall safety database and immunogenicity data for V114 to support initial licensure in adults.

ELIGIBILITY:
Inclusion Criteria:

* In good health. Any underlying chronic illness must be documented to be in stable condition.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies: a) not a woman of childbearing potential (WOCBP) OR b) a WOCBP who agrees to use 1 of the contraceptive methods as defined in the protocol during the treatment period and for at least 6 weeks after the last dose of study intervention.

Exclusion Criteria:

* History of invasive pneumococcal disease (IPD, positive blood culture, positive cerebrospinal fluid culture, or positive culture at another sterile site) or known history of other culture-positive pneumococcal disease within 3 years before Visit 1 (Day 1)
* Known hypersensitivity to any component of pneumococcal polysaccharide vaccine, pneumococcal conjugate vaccine (PCV), or any diphtheria toxoid-containing vaccine
* Known hypersensitivity to any component of influenza vaccines, including egg protein, or following a previous dose of any influenza vaccine.
* Known or suspected impairment of immunological function
* Experienced Guillain-Barré syndrome within 6 weeks of receiving a previous influenza vaccination
* Coagulation disorder contraindicating intramuscular vaccinations.
* History of malignancy ≤5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* A WOCBP who has a positive urine or serum pregnancy test before the first vaccination at Visit 1 (Day 1)
* Prior administration of any PCV (e.g., Prevnar 13®) or is expected to receive any pneumococcal vaccine during the study outside of the protocol.
* Prior administration of PNEUMOVAX®23 ≤12 months before Visit 1 (Note: individuals who received PNEUMOVAX®23 >12 months prior to Visit 1 are eligible for this study.)
* Previous receipt of influenza vaccine during the 2018/2019 flu season or expected to receive any influenza vaccine during the study outside of the protocol
* Received systemic corticosteroids (≥20 mg/day prednisone equivalent) for ≥14 consecutive days and has not completed intervention at least 30 days before study entry.
* Received systemic corticosteroids exceeding physiologic replacement doses (approximately 5 mg/day prednisone equivalent) within 14 days before vaccination (Note: Topical, ophthalmic, intra-articular or soft-tissue [e.g., bursa, tendon steroid injections], and inhaled/nebulized steroids are permitted).
* Receiving immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease
* Received a blood transfusion or blood products, including immunoglobulin within the 6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product within 30 days of receipt of study vaccine. Autologous blood transfusions are not considered an exclusion criterion.
* Is currently participating in or has participated in an interventional clinical study with an investigational compound or device within 2 months of participating in this current study.
* Is a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence as assessed by the study investigator.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (45):
- United States (45):
  - Achieve Clinical Research, LLC ( Site 0046), Birmingham, Alabama
  - Synexus Clinical Research US, Inc. ( Site 0039), Chandler, Arizona
  - Synexus Clinical Research, US,Inc/Central Arizona Medical Associates, PC ( Site 0004), Mesa, Arizona
  - Synexus Clinical Research US, Inc. ( Site 0042), Scottsdale, Arizona
  - Southland Clinical Research Center ( Site 0033), Fountain Valley, California
  - Valley Clinical Trials Inc. ( Site 0001), Northridge, California
  - Center for Clinical Trials, LLC ( Site 0025), Paramount, California
  - Artemis Institute for Clinical Research ( Site 0026), San Diego, California
  - California Research Foundation ( Site 0002), San Diego, California
  - Bayview Research Group, LLC ( Site 0010), Valley Village, California
  - Synexus Clinical Research US, Inc./Colorado Springs Family Practice ( Site 0021), Colorado Springs, Colorado
  - Indago Research & Health Center, Inc ( Site 0007), Hialeah, Florida
  - Research Centers of America, LLC ( Site 0036), Hollywood, Florida
  - Suncoast Research Group, LLC ( Site 0020), Miami, Florida
  - L&C Professional Medical Research Institute ( Site 0015), Miami, Florida
  - Alpha Science Research ( Site 0018), Miami, Florida
  - Lakes Research LLC ( Site 0034), Miami Lakes, Florida
  - Evanston Premier Healthcare & Research, LLC. ( Site 0012), Evanston, Illinois
  - Healthcare Research Network LLC ( Site 0006), Flossmoor, Illinois
  - Springfield Clinic ( Site 0045), Springfield, Illinois
  - Heartland Research Associates, LLC ( Site 0031), Augusta, Kansas
  - Heartland Research Associates, LLC ( Site 0016), Newton, Kansas
  - Kentucky Pediatric/Adult Research Inc ( Site 0011), Bardstown, Kentucky
  - Community Clinical Research Network (Marlboro, MA) ( Site 0030), Marlborough, Massachusetts
  - Healthcare Research Network LLC ( Site 0032), Hazelwood, Missouri
  - Clinical Research Center of Neveda, LLC. ( Site 0022), Las Vegas, Nevada
  - Southwest CARE Center ( Site 0013), Santa Fe, New Mexico
  - Regional Clinical Research, Inc. ( Site 0029), Endwell, New York
  - Mid Hudson Medical Research ( Site 0024), New Windsor, New York
  - Rochester Clinical Research, Inc. ( Site 0009), Rochester, New York
  - PMG Research Of Cary LLC ( Site 0035), Cary, North Carolina
  - Unity Clinical Research ( Site 0044), Lindsay, Oklahoma
  - Clinical Research Center Of Reading LLP ( Site 0014), Wyomissing, Pennsylvania
  - Omega Medical Research ( Site 0049), Warwick, Rhode Island
  - PMG Research Inc ( Site 0027), Mt. Pleasant, South Carolina
  - Holston Medical Group ( Site 0003), Bristol, Tennessee
  - Holston Medical Group ( Site 0028), Kingsport, Tennessee
  - Clinical Research Associates Inc. ( Site 0040), Nashville, Tennessee
  - Wellness Clinical Research Associates ( Site 0048), Allen, Texas
  - Benchmark Research ( Site 0037), Fort Worth, Texas
  - San Gabriel Clinical Research ( Site 0047), Georgetown, Texas
  - Synexus Clinical Research US, Inc. ( Site 0019), San Antonio, Texas
  - Charlottesville Medical Research Center, LLC ( Site 0008), Charlottesville, Virginia
  - Clinical Research Partners, LLC. ( Site 0005), Richmond, Virginia
  - Allegiance Research Specialists ( Site 0017), Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Severance R, Schwartz H, Dagan R, Connor L, Li J, Pedley A, Hartzel J, Sterling TM, Nolan KM, Tamms GM, Musey LK, Buchwald UK. Safety, tolerability, and immunogenicity of V114, a 15-valent pneumococcal conjugate vaccine, administered concomitantly with influenza vaccine in healthy adults aged >/=50 years: a randomized phase 3 trial (PNEU-FLU). Hum Vaccin Immunother. 2022 Dec 31;18(1):1-14. doi: 10.1080/21645515.2021.1976581. Epub 2021 Nov 2. PMID 34726574

RESULTS

PARTICIPANT FLOW:
Groups:
- Concomitant Group: Participants received a single 0.5 mL intramuscular (IM) injection of V114 and a single 0.5 mL IM injection of quadrivalent influenza vaccine (QIV) on Day 1 and a single 0.5 mL injection of placebo on Day 30.
- Non-Concomitant Group: Participants received a single 0.5 mL IM injection of QIV and a single 0.5 mL IM injection of placebo on Day 1 and a single 0.5 mL injection of V114 on Day 30.
Period: Overall Study
Arm/Group | Concomitant Group | Non-Concomitant Group
Started | 600 | 600
Vaccinated | 599 | 598
Completed | 583 | 583
Not Completed | 17 | 17
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 7 | 7
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 7 | 7

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study vaccination.
Groups:
- Concomitant Group: Participants received a single 0.5 mL intramuscular (IM) injection of V114 and a single 0.5 mL IM injection of QIV on Day 1 and a single 0.5 mL injection of placebo on Day 30.
- Total: Total of all reporting groups
Arm/Group | Concomitant Group | Non-Concomitant Group | Total
Number analyzed (Participants) | 599 | 598 | 1197
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (8.3) | 64.2 (8.1) | 64.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 330 | 342 | 672
  Male | 269 | 256 | 525
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 120 | 119 | 239
  Not Hispanic or Latino | 471 | 472 | 943
  Unknown or Not Reported | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 25 | 30 | 55
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 73 | 63 | 136
  White | 493 | 495 | 988
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Solicited injection-site AEs included injection-site erythema /redness, pain /tenderness, swelling.
Time Frame: Up to Day 5 after vaccination
Population: All randomized participants who received at least 1 dose of study vaccination were included. Of the 598 randomized to non-concomitant group, 1 received vaccination with concomitant group and was included (concomitant=600); 1 received 2 doses and was excluded (non-concomitant=596).
Measure: Number; unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 600 | 596
Percentage of Participants
  Injection-Site Erythema /Redness | 10.7 | 11.6
  Injection-Site Pain /Tenderness | 68.5 | 71.1
  Injection-Site Swelling | 14.2 | 16.3
Statistical Analysis 1: Comparison: Concomitant Group vs Non-Concomitant Group; Injection-Site Erythema; Test type: Other — Difference in Percent vs. Non-concomitant Group; p = 0.617, Miettinen & Nurminen; Estimated differences, confidence intervals (CIs), and p-values were calculated based on Miettinen & Nurminen method; Difference in Percent = -0.9, 95% CI 2-sided [-4.5 to 2.7]
Statistical Analysis 2: Comparison: Concomitant Group vs Non-Concomitant Group; Injection-Site Pain; Test type: Other — Difference in Percent vs. Non-concomitant Group; p = 0.320, Miettinen & Nurminen; Estimated differences, confidence intervals (CIs), and p-values were calculated based on Miettinen & Nurminen method; Difference in Percent = -2.6, 95% CI 2-sided [-7.8 to 2.6]
Statistical Analysis 3: Comparison: Concomitant Group vs Non-Concomitant Group; Injection-Site Swelling; Test type: Other — Difference in Percent vs. Non-concomitant Group; p = 0.310, Miettinen & Nurminen; Estimated differences, confidence intervals (CIs), and p-values were calculated based on Miettinen & Nurminen method; Difference in Percent = -2.1, 95% CI 2-sided [-6.2 to 2.0]

2. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Solicited systemic AEs included myalgia/muscle pain, arthralgia/joint pain, headache, and fatigue/tiredness.
Time Frame: Up to Day 14 after any vaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 600 | 596
Percentage of Participants
  Joint Pain /Arthralgia | 9.3 | 11.6
  Tiredness/Fatigue | 27.2 | 30.0
  Headache | 21.5 | 23.7
  Muscle Pain /Myalgia | 23.7 | 21.3
Statistical Analysis 1: Comparison: Concomitant Group vs Non-Concomitant Group; Arthralgia; Test type: Other — Difference in Percent vs. Non-concomitant Group; p = 0.205, Miettinen & Nurminen; Estimated differences, confidence intervals (CIs), and p-values were calculated based on Miettinen & Nurminen method; Difference in Percent = -2.2, 95% CI 2-sided [-5.8 to 1.2]
Statistical Analysis 2: Comparison: Concomitant Group vs Non-Concomitant Group; Fatigue; Test type: Other — Difference in Percent vs. Non-concomitant Group; p = 0.273, Miettinen & Nurminen; Estimated differences, confidence intervals (CIs), and p-values were calculated based on Miettinen & Nurminen method; Difference in Percent = -2.9, 95% CI 2-sided [-8.0 to 2.3]
Statistical Analysis 3: Comparison: Concomitant Group vs Non-Concomitant Group; Headache; Test type: Other — Difference in Percent vs. Non-concomitant Group; p = 0.372, Miettinen & Nurminen; Estimated differences, confidence intervals (CIs), and p-values were calculated based on Miettinen & Nurminen method; Difference in Percent = -2.2, 95% CI 2-sided [-6.9 to 2.6]
Statistical Analysis 4: Comparison: Concomitant Group vs Non-Concomitant Group; Myalgia; Test type: Other — Difference in Percent vs. Non-concomitant Group; p = 0.329, Miettinen & Nurminen; Estimated differences, confidence intervals (CIs), and p-values were calculated based on Miettinen & Nurminen method; Difference in Percent = 2.4, 95% CI 2-sided [-2.4 to 7.1]

3. Primary Outcome: Percentage of Participants With a Vaccine-Related Serious Adverse Event
Description: A serious adverse event (SAE) is an AE that results in death, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine was determined by the investigator.
Time Frame: Up to 7 months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 600 | 596
Percentage of Participants | 0 | 0
Statistical Analysis 1: Comparison: Concomitant Group vs Non-Concomitant Group; Test type: Other; Difference in Percent = 0.0, 95% CI 2-sided [-0.6 to 0.6]

4. Primary Outcome: Geometric Mean Titer (GMT) Ratio of Pneumococcal Serotype-specific Opsonophagocytic Activity (OPA)
Description: Serotype-specific OPA GMTs (estimated) and GMT ratios with 95% confidence intervals (CIs) and 1-sided p-values were calculated using a constrained longitudinal data analysis (cLDA) method utilizing data from both vaccination groups. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the GMT ratios); within-group CIs were not calculated.
Time Frame: 30 days after V114 vaccination (Day 30 for concomitant vaccination group and Day 60 for non-concomitant vaccination group)
Population: The analysis population consisted of all randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity analyses and had data available for this endpoint.
Measure: Number; unit: Titers
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 599 | 598
Titers
  Serotype 1: number analyzed (Participants) | 593 | 567
  Serotype 1 | 140.1 | 211.5
  Serotype 3: number analyzed (Participants) | 591 | 566
  Serotype 3 | 137.9 | 147.4
  Serotype 4: number analyzed (Participants) | 591 | 561
  Serotype 4 | 901.3 | 1078.5
  Serotype 5: number analyzed (Participants) | 593 | 567
  Serotype 5 | 396.1 | 500.6
  Serotype 6A: number analyzed (Participants) | 581 | 561
  Serotype 6A | 5564.2 | 6615.9
  Serotype 6B: number analyzed (Participants) | 585 | 563
  Serotype 6B | 3904.0 | 4436.5
  Serotype 7F: number analyzed (Participants) | 588 | 560
  Serotype 7F | 3563.2 | 4119.5
  Serotype 9V: number analyzed (Participants) | 591 | 566
  Serotype 9V | 2859.6 | 2874.1
  Serotype 14: number analyzed (Participants) | 589 | 567
  Serotype 14 | 2024.8 | 2228.6
  Serotype 18C: number analyzed (Participants) | 591 | 566
  Serotype 18C | 3022.8 | 3802.7
  Serotype 19A: number analyzed (Participants) | 589 | 564
  Serotype 19A | 3208.4 | 3849.0
  Serotype 19F: number analyzed (Participants) | 591 | 566
  Serotype 19F | 2523.2 | 2473.9
  Serotype 22F: number analyzed (Participants) | 586 | 560
  Serotype 22F | 2243.4 | 2932.5
  Serotype 23F: number analyzed (Participants) | 584 | 556
  Serotype 23F | 2206.2 | 2592.2
  Serotype 33F: number analyzed (Participants) | 592 | 567
  Serotype 33F | 8142.9 | 9807.4
Statistical Analysis 1: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 1; Test type: Non-Inferiority — Non-inferiority is based on the lower bound of the 95% confidence interval (CI) on the estimated GMT ratio (Concomitant Group/Nonconcomitant Group) being >0.5 (one-sided p-value < 0.025); p = 0.004, cLDA; GMT ratio, 95% CI and p-value were estimated from a constrained longitudinal data analysis (cLDA) model including all vaccinated participants; GMT Ratio = 0.66, 95% CI 2-sided [0.54 to 0.82]
Statistical Analysis 2: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.94, 95% CI 2-sided [0.81 to 1.09]
Statistical Analysis 3: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.84, 95% CI 2-sided [0.69 to 1.01]
Statistical Analysis 4: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 5; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.79, 95% CI 2-sided [0.64 to 0.98]
Statistical Analysis 5: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 6A; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.84, 95% CI 2-sided [0.71 to 1.00]
Statistical Analysis 6: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.88, 95% CI 2-sided [0.74 to 1.04]
Statistical Analysis 7: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.86, 95% CI 2-sided [0.75 to 0.99]
Statistical Analysis 8: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.99, 95% CI 2-sided [0.86 to 1.15]
Statistical Analysis 9: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 14; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.91, 95% CI 2-sided [0.77 to 1.08]
Statistical Analysis 10: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.79, 95% CI 2-sided [0.68 to 0.92]
Statistical Analysis 11: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 19A; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.83, 95% CI 2-sided [0.73 to 0.95]
Statistical Analysis 12: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 1.02, 95% CI 2-sided [0.89 to 1.17]
Statistical Analysis 13: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 22F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.77, 95% CI 2-sided [0.64 to 0.91]
Statistical Analysis 14: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.85, 95% CI 2-sided [0.70 to 1.03]
Statistical Analysis 15: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 33F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.83, 95% CI 2-sided [0.72 to 0.96]

5. Primary Outcome: GMT of Influenza Strain-Specific Hemagglutination Inhibition
Description: Activity for the 4 strains contained in QIV vaccine was determined using an hemagglutination inhibition (HAI) assay. Serotype-specific HAI GMTs (estimated) and GMT ratios with 95% confidence intervals (CIs) and 1-sided p-values were calculated using a constrained longitudinal data analysis (cLDA) method utilizing data from both vaccination groups. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the GMT ratios); within-group CIs were not calculated.
Time Frame: Day 30
Population: as for outcome 4
Measure: Number; unit: Titers
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 599 | 598
Titers
  H1N1: number analyzed (Participants) | 592 | 593
  H1N1 | 124.82 | 115.00
  H3N2: number analyzed (Participants) | 592 | 593
  H3N2 | 87.85 | 85.62
  B-Victoria: number analyzed (Participants) | 592 | 593
  B-Victoria | 35.53 | 36.88
  B-Yamagata: number analyzed (Participants) | 592 | 593
  B-Yamagata | 33.47 | 33.13
Statistical Analysis 1: Comparison: Concomitant Group vs Non-Concomitant Group; H1N1; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 1.09, 95% CI 2-sided [0.94 to 1.25]
Statistical Analysis 2: Comparison: Concomitant Group vs Non-Concomitant Group; H3N2; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 1.03, 95% CI 2-sided [0.90 to 1.17]
Statistical Analysis 3: Comparison: Concomitant Group vs Non-Concomitant Group; B-Victoria; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 0.96, 95% CI 2-sided [0.86 to 1.08]
Statistical Analysis 4: Comparison: Concomitant Group vs Non-Concomitant Group; B-Yamagata; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI and p-value were estimated from a cLDA model; GMT Ratio = 1.01, 95% CI 2-sided [0.90 to 1.13]

6. Secondary Outcome: Geometric Mean Concentration (GMC) of Pneumococcal Serotype-specific Immunoglobulin G (IgG)
Description: Serotype-specific IgG GMC ratios (estimated) and GMC ratios with 95% confidence intervals (CIs) were calculated using a constrained longitudinal data analysis (cLDA) method utilizing data from both vaccination groups. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the GMC ratios); within-group CIs were not calculated.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: µg/mL
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 599 | 598
µg/mL
  Serotype 1: number analyzed (Participants) | 592 | 568
  Serotype 1 | 4.19 | 5.41
  Serotype 3: number analyzed (Participants) | 592 | 568
  Serotype 3 | 0.75 | 0.86
  Serotype 4: number analyzed (Participants) | 592 | 568
  Serotype 4 | 1.47 | 1.86
  Serotype 5: number analyzed (Participants) | 592 | 568
  Serotype 5 | 4.65 | 5.23
  Serotype 6A: number analyzed (Participants) | 592 | 568
  Serotype 6A | 6.07 | 8.29
  Serotype 6B: number analyzed (Participants) | 592 | 568
  Serotype 6B | 7.11 | 9.26
  Serotype 7F: number analyzed (Participants) | 592 | 568
  Serotype 7F | 4.68 | 5.33
  Serotype 9V: number analyzed (Participants) | 592 | 568
  Serotype 9V | 3.84 | 4.26
  Serotype 14: number analyzed (Participants) | 592 | 568
  Serotype 14 | 8.30 | 9.80
  Serotype 18C: number analyzed (Participants) | 592 | 568
  Serotype 18C | 9.99 | 12.75
  Serotype 19A: number analyzed (Participants) | 592 | 568
  Serotype 19A | 13.43 | 15.09
  Serotype 19F: number analyzed (Participants) | 592 | 568
  Serotype 19F | 8.68 | 9.75
  Serotype 22F: number analyzed (Participants) | 592 | 568
  Serotype 22F | 3.29 | 4.33
  Serotype 23F: number analyzed (Participants) | 592 | 568
  Serotype 23F | 5.68 | 6.82
  Serotype 33F: number analyzed (Participants) | 592 | 568
  Serotype 33F | 9.19 | 10.69
Statistical Analysis 1: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 1; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.77, 95% CI 2-sided [0.67 to 0.89]
Statistical Analysis 2: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 3; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.87, 95% CI 2-sided [0.76 to 0.99]
Statistical Analysis 3: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 4; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.79, 95% CI 2-sided [0.68 to 0.91]
Statistical Analysis 4: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 5; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.89, 95% CI 2-sided [0.77 to 1.02]
Statistical Analysis 5: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 6A; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.73, 95% CI 2-sided [0.61 to 0.87]
Statistical Analysis 6: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 6B; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.77, 95% CI 2-sided [0.64 to 0.91]
Statistical Analysis 7: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 7F; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.88, 95% CI 2-sided [0.76 to 1.01]
Statistical Analysis 8: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 9V; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.90, 95% CI 2-sided [0.79 to 1.03]
Statistical Analysis 9: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 14; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.85, 95% CI 2-sided [0.73 to 0.99]
Statistical Analysis 10: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 18C; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.78, 95% CI 2-sided [0.68 to 0.91]
Statistical Analysis 11: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 19A; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.89, 95% CI 2-sided [0.78 to 1.02]
Statistical Analysis 12: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 19F; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.89, 95% CI 2-sided [0.77 to 1.03]
Statistical Analysis 13: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 22F; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.76, 95% CI 2-sided [0.65 to 0.89]
Statistical Analysis 14: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 23F; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.83, 95% CI 2-sided [0.70 to 0.98]
Statistical Analysis 15: Comparison: Concomitant Group vs Non-Concomitant Group; Serotype 33F; Test type: Other — GMC ratio and 95% CI were estimated from cLDA model; GMC Ratio = 0.86, 95% CI 2-sided [0.75 to 0.99]

7. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Pneumococcal Serotype-Specific OPA
Description: Activity for the 15 serotypes contained in V114 vaccine will be determined using a Multiplex Opsonophagocytic Assay. GMFR is the geometric mean of fold rise from baseline to postvaccination.
Time Frame: Baseline and 30 days after V114 vaccination (Day 1 and Day 30 for concomitant vaccination group, and Day 30 and Day 60 for non-concomitant vaccination group, respectively)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 599 | 598
Ratio
  Serotype 1: number analyzed (Participants) | 517 | 505
  Serotype 1 | 8.0 [6.8 to 9.3] | 11.8 [10.1 to 13.9]
  Serotype 3: number analyzed (Participants) | 495 | 493
  Serotype 3 | 4.7 [4.3 to 5.3] | 4.8 [4.3 to 5.4]
  Serotype 4: number analyzed (Participants) | 471 | 476
  Serotype 4 | 9.4 [8.0 to 11.0] | 11.5 [9.7 to 13.6]
  Serotype 5: number analyzed (Participants) | 516 | 503
  Serotype 5 | 8.1 [7.0 to 9.4] | 10.2 [8.7 to 12.0]
  Serotype 6A: number analyzed (Participants) | 443 | 451
  Serotype 6A | 10.5 [9.1 to 12.1] | 12.1 [10.5 to 14.0]
  Serotype 6B: number analyzed (Participants) | 466 | 481
  Serotype 6B | 17.6 [14.8 to 20.9] | 20.5 [17.3 to 24.4]
  Serotype 7F: number analyzed (Participants) | 492 | 484
  Serotype 7F | 9.2 [7.9 to 10.8] | 8.0 [6.9 to 9.4]
  Serotype 9V: number analyzed (Participants) | 483 | 483
  Serotype 9V | 5.8 [5.1 to 6.6] | 5.3 [4.6 to 6.1]
  Serotype 14: number analyzed (Participants) | 498 | 491
  Serotype 14 | 3.9 [3.3 to 4.4] | 4.1 [3.5 to 4.7]
  Serotype 18C: number analyzed (Participants) | 503 | 491
  Serotype 18C | 9.8 [8.6 to 11.2] | 11.6 [10.0 to 13.4]
  Serotype 19A: number analyzed (Participants) | 482 | 476
  Serotype 19A | 6.2 [5.4 to 7.2] | 6.6 [5.7 to 7.6]
  Serotype 19F: number analyzed (Participants) | 490 | 492
  Serotype 19F | 5.2 [4.6 to 5.9] | 4.7 [4.2 to 5.4]
  Serotype 22F: number analyzed (Participants) | 438 | 446
  Serotype 22F | 15.9 [12.8 to 19.8] | 20.6 [16.4 to 25.9]
  Serotype 23F: number analyzed (Participants) | 427 | 436
  Serotype 23F | 13.9 [11.7 to 16.6] | 11.9 [9.9 to 14.3]
  Serotype 33F: number analyzed (Participants) | 510 | 488
  Serotype 33F | 4.3 [3.8 to 4.9] | 4.6 [4.0 to 5.3]

8. Secondary Outcome: GMFR in Pneumococcal Serotype-Specific IgG
Description: Immunoglobulin G for the 15 serotypes contained in V114 vaccine will be determined using an electrochemiluminescence assay. GMFR is the geometric mean of fold rise from baseline to postvaccination.
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 599 | 598
Ratio
  Serotype 1: number analyzed (Participants) | 568 | 549
  Serotype 1 | 6.1 [5.5 to 6.9] | 7.5 [6.6 to 8.5]
  Serotype 3: number analyzed (Participants) | 568 | 549
  Serotype 3 | 4.4 [4.0 to 4.8] | 5.1 [4.6 to 5.7]
  Serotype 4: number analyzed (Participants) | 568 | 549
  Serotype 4 | 5.3 [4.8 to 5.9] | 6.5 [5.8 to 7.4]
  Serotype 5: number analyzed (Participants) | 568 | 550
  Serotype 5 | 3.5 [3.2 to 3.9] | 4.0 [3.5 to 4.5]
  Serotype 6A: number analyzed (Participants) | 568 | 549
  Serotype 6A | 15.6 [13.7 to 17.8] | 19.9 [17.3 to 22.9]
  Serotype 6B: number analyzed (Participants) | 566 | 549
  Serotype 6B | 14.0 [12.2 to 15.9] | 17.8 [15.5 to 20.5]
  Serotype 7F: number analyzed (Participants) | 568 | 550
  Serotype 7F | 6.7 [6.0 to 7.5] | 7.2 [6.4 to 8.2]
  Serotype 9V: number analyzed (Participants) | 568 | 547
  Serotype 9V | 5.9 [5.3 to 6.6] | 6.6 [5.8 to 7.4]
  Serotype 14: number analyzed (Participants) | 568 | 549
  Serotype 14 | 3.8 [3.4 to 4.3] | 4.4 [3.9 to 5.0]
  Serotype 18C: number analyzed (Participants) | 567 | 549
  Serotype 18C | 11.2 [9.8 to 12.8] | 12.9 [11.2 to 14.9]
  Serotype 19A: number analyzed (Participants) | 567 | 549
  Serotype 19A | 6.4 [5.7 to 7.1] | 6.8 [6.1 to 7.7]
  Serotype 19F: number analyzed (Participants) | 567 | 549
  Serotype 19F | 8.1 [7.2 to 9.2] | 8.9 [7.9 to 10.1]
  Serotype 22F: number analyzed (Participants) | 568 | 550
  Serotype 22F | 7.6 [6.6 to 8.6] | 10.1 [8.8 to 11.6]
  Serotype 23F: number analyzed (Participants) | 568 | 548
  Serotype 23F | 10.7 [9.4 to 12.2] | 11.9 [10.3 to 13.7]
  Serotype 33F: number analyzed (Participants) | 568 | 549
  Serotype 33F | 5.5 [4.8 to 6.1] | 6.0 [5.3 to 6.8]

9. Secondary Outcome: Percentage of Participants With GMFR ≥4 in Pneumococcal Serotype-specific OPA
Description: Activity for the 15 serotypes contained in V114 vaccine will be determined using a Multiplex Opsonophagocytic Assay. GMFR is the geometric mean of fold rise from baseline to postvaccination. The percentage of participants who had ≥ 4-fold rise in GMFR were calculated from baseline to postvaccination.
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 599 | 598
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 517 | 505
  Serotype 1 | 57.8 [53.4 to 62.1] | 66.3 [62.0 to 70.5]
  Serotype 3: number analyzed (Participants) | 495 | 493
  Serotype 3 | 54.7 [50.2 to 59.2] | 54.8 [50.3 to 59.2]
  Serotype 4: number analyzed (Participants) | 471 | 476
  Serotype 4 | 63.1 [58.5 to 67.4] | 66.4 [61.9 to 70.6]
  Serotype 5: number analyzed (Participants) | 516 | 503
  Serotype 5 | 60.5 [56.1 to 64.7] | 63.4 [59.0 to 67.6]
  Serotype 6A: number analyzed (Participants) | 443 | 451
  Serotype 6A | 71.1 [66.6 to 75.3] | 75.6 [71.4 to 79.5]
  Serotype 6B: number analyzed (Participants) | 466 | 481
  Serotype 6B | 72.5 [68.2 to 76.5] | 76.1 [72.0 to 79.8]
  Serotype 7F: number analyzed (Participants) | 492 | 484
  Serotype 7F | 63.0 [58.6 to 67.3] | 59.7 [55.2 to 64.1]
  Serotype 9V: number analyzed (Participants) | 483 | 483
  Serotype 9V | 54.9 [50.3 to 59.4] | 53.4 [48.9 to 57.9]
  Serotype 14: number analyzed (Participants) | 498 | 491
  Serotype 14 | 38.6 [34.3 to 43.0] | 40.9 [36.6 to 45.4]
  Serotype 18C: number analyzed (Participants) | 503 | 491
  Serotype 18C | 67.4 [63.1 to 71.5] | 70.3 [66.0 to 74.3]
  Serotype 19A: number analyzed (Participants) | 482 | 476
  Serotype 19A | 53.7 [49.2 to 58.3] | 57.1 [52.6 to 61.6]
  Serotype 19F: number analyzed (Participants) | 490 | 492
  Serotype 19F | 53.7 [49.1 to 58.2] | 48.8 [44.3 to 53.3]
  Serotype 22F: number analyzed (Participants) | 438 | 446
  Serotype 22F | 64.2 [59.5 to 68.7] | 67.5 [62.9 to 71.8]
  Serotype 23F: number analyzed (Participants) | 427 | 436
  Serotype 23F | 73.1 [68.6 to 77.2] | 67.2 [62.6 to 71.6]
  Serotype 33F: number analyzed (Participants) | 510 | 488
  Serotype 33F | 44.1 [39.8 to 48.5] | 44.9 [40.4 to 49.4]

10. Secondary Outcome: Percentage of Participants With GMFR ≥4 in Pneumococcal Serotype-specific IgG
Description: Immunoglobulin G for the 15 serotypes contained in V114 vaccine will be determined using an electrochemiluminescence assay. GMFR is the geometric mean of fold rise from baseline to postvaccination. The percentage of participants who had ≥ 4-fold rise in GMFR are calculated from baseline to postvaccination.
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 599 | 598
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 568 | 549
  Serotype 1 | 54.8 [50.6 to 58.9] | 60.8 [56.6 to 64.9]
  Serotype 3: number analyzed (Participants) | 568 | 549
  Serotype 3 | 46.8 [42.7 to 51.0] | 50.6 [46.4 to 54.9]
  Serotype 4: number analyzed (Participants) | 568 | 549
  Serotype 4 | 53.7 [49.5 to 57.9] | 57.2 [52.9 to 61.4]
  Serotype 5: number analyzed (Participants) | 568 | 550
  Serotype 5 | 38.0 [34.0 to 42.2] | 40.4 [36.2 to 44.6]
  Serotype 6A: number analyzed (Participants) | 568 | 549
  Serotype 6A | 77.3 [73.6 to 80.7] | 79.2 [75.6 to 82.6]
  Serotype 6B: number analyzed (Participants) | 566 | 549
  Serotype 6B | 74.9 [71.1 to 78.4] | 79.1 [75.4 to 82.4]
  Serotype 7F: number analyzed (Participants) | 568 | 550
  Serotype 7F | 60.2 [56.1 to 64.3] | 59.6 [55.4 to 63.8]
  Serotype 9V: number analyzed (Participants) | 568 | 547
  Serotype 9V | 54.4 [50.2 to 58.6] | 55.4 [51.1 to 59.6]
  Serotype 14: number analyzed (Participants) | 568 | 549
  Serotype 14 | 39.8 [35.7 to 43.9] | 43.0 [38.8 to 47.2]
  Serotype 18C: number analyzed (Participants) | 567 | 549
  Serotype 18C | 67.5 [63.5 to 71.4] | 68.9 [64.8 to 72.7]
  Serotype 19A: number analyzed (Participants) | 567 | 549
  Serotype 19A | 59.3 [55.1 to 63.3] | 60.1 [55.9 to 64.2]
  Serotype 19F: number analyzed (Participants) | 567 | 549
  Serotype 19F | 63.7 [59.6 to 67.6] | 66.7 [62.6 to 70.6]
  Serotype 22F: number analyzed (Participants) | 568 | 550
  Serotype 22F | 56.5 [52.3 to 60.6] | 64.9 [60.8 to 68.9]
  Serotype 23F: number analyzed (Participants) | 568 | 548
  Serotype 23F | 67.4 [63.4 to 71.3] | 69.7 [65.7 to 73.5]
  Serotype 33F: number analyzed (Participants) | 568 | 549
  Serotype 33F | 50.4 [46.2 to 54.5] | 53.9 [49.6 to 58.1]

11. Secondary Outcome: GMFR of Influenza Strain-Specific HAI
Description: Activity for the 4 strains contained in QIV vaccine will be determined using an HAI assay. GMFR is the geometric mean of fold rise from baseline to postvaccination.
Time Frame: Baseline (Day 1) and Day 30
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 599 | 598
Ratio
  H1N1: number analyzed (Participants) | 569 | 561
  H1N1 | 4.2 [3.8 to 4.7] | 4.2 [3.8 to 4.8]
  H3N2: number analyzed (Participants) | 569 | 561
  H3N2 | 2.2 [2.0 to 2.4] | 2.2 [2.0 to 2.4]
  B-Victoria: number analyzed (Participants) | 569 | 561
  B-Victoria | 2.1 [2.0 to 2.3] | 2.2 [2.0 to 2.4]
  B-Yamagata: number analyzed (Participants) | 569 | 561
  B-Yamagata | 2.3 [2.1 to 2.5] | 2.3 [2.1 to 2.4]

12. Secondary Outcome: Percentage of Participants With Influenza Strain-specific HAI Titer ≥1:40
Description: Activity for the 4 strains contained in QIV vaccine will be determined using an HAI assay. Seroconversion is defined as achieving a 4-fold rise from baseline to postvaccination among participants who are seropositive at baseline (HAI titer ≥ 1:10) or a titer of ≥ 1:40 at postvaccination among participants who are seronegative at baseline (HAI titer < 1:10).
Time Frame: Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 599 | 598
Percentage of Participants
  H1N1: number analyzed (Participants) | 576 | 567
  H1N1 | 85.9 [82.8 to 88.7] | 84.7 [81.4 to 87.5]
  H3N2: number analyzed (Participants) | 576 | 567
  H3N2 | 77.4 [73.8 to 80.8] | 79.2 [75.6 to 82.5]
  B-Victoria: number analyzed (Participants) | 576 | 567
  B-Victoria | 55.0 [50.9 to 59.1] | 54.9 [50.6 to 59.0]
  B-Yamagata: number analyzed (Participants) | 576 | 567
  B-Yamagata | 52.4 [48.3 to 56.6] | 50.8 [46.6 to 55]

13. Secondary Outcome: Percentage of Participants Who Seroconvert for Influenza Strain-specific HAI
Description: Activity for the 4 strains contained in QIV vaccine will be determined using an HAI assay. Seroconversion for HAI responses is defined as achieving either 1) a 4-fold rise in influenza strain-specific HAI titer from Baseline to Day 30 among participants who are seropositive at Baseline (HAI titer ≥1:10) or 2) a influenza strain-specific HAI titer of ≥1:40 at Day 30 among participants who are seronegative at Baseline (HAI titer <1:10).
Time Frame: Baseline (Day 1) and Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Concomitant Group | Non-Concomitant Group
Number analyzed (Participants) | 599 | 598
Percentage of Participants
  H1N1: number analyzed (Participants) | 569 | 561
  H1N1 | 48.5 [44.3 to 52.7] | 48.3 [44.1 to 52.5]
  H3N2: number analyzed (Participants) | 569 | 561
  H3N2 | 27.8 [24.1 to 31.6] | 25.3 [21.8 to 29.1]
  B-Victoria: number analyzed (Participants) | 569 | 561
  B-Victoria | 29.2 [25.5 to 33.1] | 28.7 [25.0 to 32.6]
  B-Yamagata: number analyzed (Participants) | 569 | 561
  B-Yamagata | 31.1 [27.3 to 35.1] | 30.5 [26.7 to 34.5]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected up to 14 days following each vaccination. Serious adverse events and all-cause mortality were reported throughout the duration of the study, up to 7 months.
Description: The analysis population consisted of all randomized participants who received at least 1 dose of study vaccination. Of 598 participants randomized to non-concomitant group, 1 participant received vaccination with concomitant group and was included for safety analyses (concomitant=600); 1 participant received V114 at both vaccination visits and was excluded from the safety analyses (non-concomitant=596). The all-cause mortality was assessed in all randomized participants.
Groups:
- Concomitant Group (V114, QIV, Placebo): Participants received a single 0.5 mL intramuscular (IM) injection of V114 and a single 0.5 mL IM injection of QIV on Day 1 and a single 0.5 mL injection of placebo on Day 30.
- Noncomitant Group (Placebo, QIV, V114): Participants received a single 0.5 mL IM injection of QIV and a single 0.5 mL IM injection of placebo on Day 1 and a single 0.5 mL injection of V114 on Day 30.
Arm/Group | Concomitant Group (V114, QIV, Placebo) | Noncomitant Group (Placebo, QIV, V114)
All-Cause Mortality (participants affected / at risk) | 1/600 | 0/600
Serious Adverse Events (participants affected / at risk) | 22/600 | 14/596
Other Adverse Events (participants affected / at risk) | 458/600 | 473/596
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Group (V114, QIV, Placebo) (N=600) | Noncomitant Group (Placebo, QIV, V114) (N=596)
Cardiac failure congestive (Cardiac disorders) | 3 (4) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Group (V114, QIV, Placebo) (N=600) | Noncomitant Group (Placebo, QIV, V114) (N=596)
Fatigue (General disorders) | 163 (242) | 179 (274)
Injection site erythema (General disorders) | 65 (94) | 70 (87)
Injection site pain (General disorders) | 413 (684) | 424 (710)
Injection site swelling (General disorders) | 86 (124) | 99 (128)
Arthralgia (Musculoskeletal and connective tissue disorders) | 56 (69) | 69 (88)
Myalgia (Musculoskeletal and connective tissue disorders) | 142 (180) | 127 (154)
Headache (Nervous system disorders) | 129 (183) | 143 (215)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03615482/Prot_SAP_000.pdf